CLINICAL TRIAL: NCT03104062
Title: Effect of Ticagrelor and Clopidogrel on Coronary Microcirculation in Patients With Acute Myocardial Infarction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Marco Antonio Scanavini Filho, Principal Investigator, University of Sao Paulo General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 4416
Record Dates: First submitted 2017-03-17; First posted 2017-04-07 (Actual); Last update posted 2018-05-18 (Actual); Status verified 2018-05

CONDITIONS: Coronary Microvascular Disease; Ticagrelor; Thrombolysis; Microbubble Contrasted Echocardiography
MeSH Terms: conditions — Microvascular Angina

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ticagrelor (Other): Patients will be randomized to have Ticagrelor 90mg BID
  Interventions: Diagnostic Test: Microbubble Contrasted Echocardiography; Diagnostic Test: Platelet Aggregability; Diagnostic Test: Laboratory
- Clopidogrel (Other): Patientes will be randomized to have Clopidogrel 75mg once a day
  Interventions: Diagnostic Test: Microbubble Contrasted Echocardiography; Diagnostic Test: Platelet Aggregability; Diagnostic Test: Laboratory

INTERVENTIONS:
Diagnostic Test: Microbubble Contrasted Echocardiography — Myocardial Perfusion Score Index (MPSI) obtained using Microbubble Contrasted Echocardiography
Diagnostic Test: Platelet Aggregability — Obtained using Multiplate Analyzer
Diagnostic Test: Laboratory — it will be collected at patients arrival, Reative C-Protein, BNP, CK-mass, Troponine, interleukine-6, Creatinine.

SUMMARY:
Of the patients diagnosed with ST-segment elevation myocardial infarction (STEMI) who underwent reperfusion therapy and have thrombolysis in myocardial infarction (TIMI) 3 flow, about 40% have flow alterations in the coronary microcirculation, which leads to worse remodeling of the left ventricle with a consequent increase in the mortality of this population. Clopidogrel is the only known antiplatelet medication that brings benefits to the coronary microcirculation. Ticagrelor is significantly superior to clopidogrel in terms of decreasing mortality.

The main objective of this study is to compare the effect of ticagrelor versus clopidogrel on the coronary microcirculation by the Myocardial Perfusion Score Index (MPSI) obtained using Microbubble Contrasted Echocardiography (MCE) in patients who have STEMI and treated with thrombolysis.

DETAILED DESCRIPTION:
The present project should prospectively include patients participating in the TREAT study, who are including individuals with Acute Myocardial Infarction (AMI) treated with fibrinolytic and openly randomized to ticagrelor or clopidogrel within 24 hours of the onset of symptoms. Patients will be submitted to coronary angiography within 4 (± 2) days of the onset of symptoms, and those who, at the end of coronary angiography, present residual obstruction in the culprit vessel of less than 50% and have TIMI 3 flow, regardless of have undergone percutaneous coronary intervention will be included.

Following, on day 2 (± 1) days after coronary angiography (therefore 6 ± 3 days from the onset of symptoms), they will be submitted to microcirculation perfusion evaluation by means of MPSI (myocardial perfusion score index) obtained by MCE (Microbubble contrasted echocardiography) - blood collection for evaluation of Platelet aggregability will be performed immediately prior to the start of MCE. Finally, in order to evaluate left ventricular remodeling, patients will undergo a new Echocardiography within 90 (± 10) days after discharge.

ELIGIBILITY:
Inclusion Criteria:

* age from 18 years old to 75 years old.
* Patients with a ST-segment elevation AMI with up to 24 hours duration, documented by ischemic symptoms due to atherosclerosis> 10 minutes at rest, treated with pharmacological thrombolysis, acetylsalicylic acid (ASA) and Clopidogrel or Ticagrelor.
* Cardiac catheterization performed within 4 (± 2) days of the onset of symptoms, which at the end of coronary angiography showed residual obstruction in the "culprit" artery <50% with TIMI 3 flow regardless of whether or not the percutaneous coronary intervention was performed.

Exclusion Criteria:

* Previous infarction known from the same wall as the current one
* Any contraindication to the use of Clopidogrel or Ticagrelor
* Need for oral anticoagulation therapy or aspirin doses greater than 100mg per day.
* Concomitant oral or intravenous therapy with strong inhibitors of Cytochrome P450, family 3, subfamily A (CYP3A), Substrates of CYP3A with narrow therapeutic indices or strong inducers of CYP3A
* High risk of bradyarrhythmias
* Dialysis therapy
* Clinically important thrombocytopenia known
* Clinically Significant Anemia
* Pregnancy or lactation
* Contraindications to fibrinolytic therapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Myocardial Perfusion Score Index (MPSI) | 4 (±3) days after Cardiac catheterization
  Obtained using Microbubble Contrasted Echocardiography

SECONDARY OUTCOMES:
Left ventricular remodeling 90 days after de AMI, using Echocargiography parameters (End diastolic volume, end systolic volume and ejection Fraction) | after 90 days after discharge
  To compare the parameters of left ventricular remodeling (End diastolic volume, End Systolic Volume, Ejection Fraction) at after 90 days after discharge from the ticagrelor and clopidogrel groups
number of myocardial segments with perfusion deficit in coronary microcirculation | 4 (±3) days after Cardiac catheterization
  To evaluate the number of myocardial segments with perfusion deficit in coronary microcirculation in the ticagrelor and clopidogrel groups
MPSI in patients submitted to angioplasty | 4 (±3) days after Cardiac catheterization
  To evaluate MPSI in the subgroups of patients submitted to angioplasty and not submitted to angioplasty
Patients who used clopidogrel prior to randomization and were randomized to ticagrelor | 4 (±3) days after Cardiac catheterization
  To evaluate MPSI in subgroups of patients who used clopidogrel prior to randomization and were randomized to ticagrelor
Elective versus Urgent Percutaneous Coronary Intervention (PCI) | 4 (±3) days after Cardiac catheterization
  To compare the ticagrelor and clopidogrel groups in patients who had elective or urgent PCI
Platelet aggregability | 4 (±3) days after Cardiac catheterization
  To evaluate the platelet aggregability in the ticagrelor and clopidogrel groups obtained immediately before Myocardial Contrasted Echocardiography (MCE) by Multiplate
Time Ticagrelor or Clopidogrel is administered | 4 (±3) days after Cardiac catheterization
  Evaluate the main objective of the study in two subgroups: 1) Ticagrelor or Clopidogrel administered less than 12 hours from the symptoms onset. 2) greater than or equal to 12 hours from the symptoms onset

OTHER OUTCOMES:
Laboratory analysis | 4 (±3) days after Cardiac catheterization
  Number of Participants With Abnormal Laboratory Values in both groups, Ticagrelor and Clopidogrel. The laboratory analysis will be: Platelet count; Platelet mean volume; HbA1C; Creatinine clearance; Reactive c-protein; Interleucine-6; Brain natriuretic peptide (BNP); Troponin; Creatine Kinase-MB (CK-MB);
In hospital use of morphine (Yes or No) | 4 (±3) days after Cardiac catheterization
  Evaluate MPSI in patients who used Morphine or not.
In hospital Use of Proton Pump Inhibitor (PPI) (yes or no) | 4 (±3) days after Cardiac catheterization
  Evaluate MPSI in patients who used PPI or not

CONTACTS AND LOCATIONS:
Locations (1):
- Heart Institute (InCor) - University of Sao Paulo Medical School, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Scanavini-Filho MA, Berwanger O, Matthias W, Aguiar MO, Chiang HP, Azevedo L, Baracioli LM, Lima FG, Furtado RHM, Dalcoquio TF, Menezes FR, Ferrari AG, de Luca F, Giugliano RP, Goodman S, Nicolau JC. Effects of Ticagrelor and Clopidogrel on Coronary Microcirculation in Patients with Acute Myocardial Infarction. Adv Ther. 2022 Apr;39(4):1832-1843. doi: 10.1007/s12325-022-02061-0. Epub 2022 Feb 26. PMID 35218519